CLINICAL TRIAL: NCT01605799
Title: A Novel PTSD Treatment for Veterans Who Killed in War
Brief Title: IOK Treatment Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RRP 12-237
Record Dates: First submitted 2012-05-18; First posted 2012-05-25 (Estimated); Results first posted 2015-12-17 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-01

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD; Mental Health; War; Veterans
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IOK Treatment (Active Comparator): Six to eight week treatment lasting one to 1.5 hours addressing maladaptive cognitions related to killing in war.
  Interventions: Behavioral: IOK Killing Treatment
- Wait list control group (Placebo Comparator): Participants in this group will not receive treatment; however, at the end of 6 weeks, they will be offered the option of receiving treatment.
  Interventions: Behavioral: IOK Killing Treatment; Behavioral: Wait list control group

INTERVENTIONS:
Behavioral: IOK Killing Treatment — The IOK Killing Treatment is based on Cognitive Behavioral Therapy theory and principals and target maladaptive cognitions related to killing in war.
Behavioral: Wait list control group — Participants in this group will not receive treatment; however, at the end of 6 weeks, they will be offered the option of receiving treatment.
  Arms: Wait list control group

SUMMARY:
The goals of this project are

* 1) to evaluate the effectiveness of a CBT treatment module addressing the mental health and functional impact of killing in the war zone,
* 2) to gather data on Veteran stakeholders' perceptions of acceptability and feasibility of the CBT treatment module, which would be used to further refine the intervention, and
* 3) to gather data on clinician stakeholders' perceptions of acceptability and feasibility of the CBT treatment module, which would be used to ensure that the module could be easily integrated into EBT for PTSD.

DETAILED DESCRIPTION:
Background: There is mounting evidence that Veterans from multiple eras who kill in war are at increased risk for posttraumatic stress disorder (PTSD), alcohol abuse, suicide, and functional difficulties after returning home. Despite high rates of exposure to killing and associated maladaptive responses, the military and VA do not routinely assess exposure to killing, which could assist with prevention and treatment efforts. Furthermore, the impact of killing is not currently addressed as a component of evidence-based treatment (EBT) for PTSD. In fact, in the current system, a Veteran can receive PTSD evaluation and evidence-based treatment without ever being asked about killing and its impact. Some researchers have cautioned against using one type of PTSD treatment, one commonly used in the VA, suggesting that it may be harmful for these patients. Consequently, it is possible that failing to directly treat the mental health impact of killing could result in inappropriate treatment, cause harm to Veterans, and cost lives.

Objectives: Our first aim is to evaluate the effectiveness of a CBT treatment module addressing the mental health and functional impact of killing in the war zone, which would be added onto existing EBT for PTSD. Our second aim is to gather data on Veteran stakeholders' perceptions of acceptability and feasibility of the CBT treatment module, which would be used to further refine the intervention. Our third aim is to gather data on clinician stakeholders' perceptions of acceptability and feasibility of the CBT treatment module, which would be used to ensure that the module could be easily integrated into EBT for PTSD.

Methods: The investigators propose a 12-month pilot, cross-sectional Hybrid Type 2 study, given that The investigators will be adding a treatment module to existing EBT for PTSD. The investigators will conduct a randomized, controlled effectiveness trial to better understand if the six-week treatment module addressing the impact of killing has added benefit, compared to PTSD treatment as usual (N = 50). The investigators will employ a concurrent design mixed method study to test the perceptions of Veteran stakeholders who receive the treatment module, obtaining ratings of acceptability and feasibility through self-report measures and interviews. The investigators also will interview clinicians who provide EBT for PTSD, and interviews will be guided by Roger's five intrinsic characteristics, as outlined in his Diffusion of Innovations Theory.

Impact: Through involving Veteran and clinician stakeholders, the main impact of this project will be to obtain information that will assist in revising the CBT treatment module and help prepare for implementing the module in already existing settings, where EBT for PTSD is provided.

ELIGIBILITY:
Inclusion Criteria:

* Combat Veterans ranging in age from 18-70 years will be recruited to participate in this study. Combat veterans ranging in age from 70 to 90 years will also be considered for enrollment in the study on a case-by-case basis.
* Veterans will need to endorse having taken a life in a war zone context, to meet criteria for PTSD, and to have received some prior treatment for PTSD to be included in the study.
* Participants in current PTSD treatment will not be excluded; however, if receiving medications, they will need to be stabilized on current medications for at least one month.
* If receiving Prolonged Exposure (PE) or Cognitive Processing Therapy (CPT), the two treatments the VA recognizes as evidence-based treatment for PTSD, individuals will need to wait two weeks after they have completed the treatment in order to enroll in the study, and new baseline measures will be obtained at that time.

Exclusion Criteria:

* Potential participants will only be excluded if they meet current or lifetime criteria for a psychotic disorder.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2012-10; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shira Maguen, PhD, Principal Investigator — San Francisco VA Medical Center, San Francisco, CA
Locations (1):
- San Francisco VA Medical Center, San Francisco, CA, San Francisco, California, United States

REFERENCES:
- [Result] Maguen S, Burkman K. Combat-Related Killing: Expanding Evidence-Based Treatments for PTSD. Cognitive and behavioral practice. 2013 Nov 1; 20(4):476-479.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IOK Treatment | Wait List Control Group
Started | 17 | 16
Completed | 15 | 15
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IOK Treatment | Wait List Control Group | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (12.8) | 60.5 (14.3) | 59.9 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 15 | 15 | 30
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1 | 0 | 1
  Black | 3 | 3 | 6
  Caucasian | 7 | 11 | 18
  Latino | 1 | 0 | 1
  Multiracial | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in PTSD Symptoms as Measured by the PCL
Description: The PCL is a 17 item self-report measure of the 17 symptoms of PTSD per the DSM IV. Possible scores range from 17 (better outcome) to 85 (worse outcome).
Time Frame: PTSD symptoms will be assessed at Baseline or the first study visit and the end of treatment (Week 7)
Population: The mean change in PCL score from baseline to end of treatment will be measured using an intent to treat analysis.
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | IOK Treatment | Wait List Control Group
Number analyzed (Participants) | 15 | 15
Units on a scale | -7.33 [-14.71 to -0.05] | -2.13 [-5.97 to -1.71]

2. Secondary Outcome: Change in Psychological Symptoms as Measured by the Brief Symptom Inventory (BSI-53)
Description: The BSI is a 53 item self-report scale used to measure nine primary symptom dimensions (somatization, obsessive-compulsive behavior, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation, and psychoticism). Respondents rank each feeling item (e.g., "your feelings being easily hurt") on a 5-point scale ranging from 0 (not at all) to 4 (extremely). Rankings characterize the intensity of distress during the past seven days. The total score is the sum of all responses [minimum = 0 (better outcome), maximum = 212 (worse outcome)].
Time Frame: The BSI will be administered at Baseline or the first study visit and the end of treatment (Week 7)
Population: The mean change in BSI between baseline and end of treatment will be measured using an intent to treat analysis.
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | IOK Treatment | Wait List Control Group
Number analyzed (Participants) | 15 | 15
Units on a scale | -17.73 [-32.87 to -2.6] | 4.53 [-6.65 to 15.71]

ADVERSE EVENTS:
Arm/Group | IOK Treatment | Wait List Control Group
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No